CLINICAL TRIAL: NCT04553302
Title: Comparison of Hand Functions and Wrist Proprioception in Patients With and Without Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Melissa Köprülüoğlu (Other)
Responsible Party: Sponsor-Investigator, Melissa Köprülüoğlu, Research Assistant, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Other Study IDs: Izmir Katip Celebi University
Record Dates: First submitted 2020-09-05; First posted 2020-09-17 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis, Hand Function, Wrist Proprioception.
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psoriatic Arthritis: Patients diagnosed with PsA according to CASPAR criteria by the rheumatologist were included.
  Interventions: Other: This study does not contain any intervention.
- Rheumatoid Arthritis: Patients diagnosed with RA according to ACR / EULAR 2010 criteria by the rheumatologist were included.
  Interventions: Other: This study does not contain any intervention.
- Asymptomatic Healthy Group: Participants had any neurological and/or rheumatological diseases, no complaints about the upper extremity. Participants diagnosed with OA according to traditional clinical criteria were excluded from the study.
  Interventions: Other: This study does not contain any intervention.

INTERVENTIONS:
Other: This study does not contain any intervention. — This study does not contain any intervention.

SUMMARY:
The purpose of this study is to assess hand functions and wrist joint position sense in patients with and without PsA.

DETAILED DESCRIPTION:
In this study, 54 patients (18 of them RA, 18 of them PsA and, 18 of them asymptomatic healthy group) were included. The patient group was selected from the patients who came to the Izmir Katip Celebi University Ataturk Training and Research Hospital Rheumatology Outpatient Clinic for routine control.

Participants were matched according to age and gender. It was recorded demographic and clinical data.

Grip and pinch strengths were evaluated within the scope of hand function evaluation. Wrist joint position sense was evaluated along with hand functions.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed according to CASPAR or ACR/ EULAR 2010 criteria for patient groups
* taking regular medication for patient groups,
* have complaints related to hand / wrist joints for patients groups,
* have no complaints related to upper extremity for asymptomatic healthy group.
* have any rheumatologic disease and OA diagnosed according to traditional criteria

Exclusion Criteria:

* finger infection and / or finger amputation,
* using orthoses,
* to report a diagnosis of neurological disease,
* to report a history of trauma or surgery involving the upper extremity,
* to report a psychiatric and / or cognitive problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 54 participants
  * 18 of them PsA
  * 18 of them RA
  * 18 of them asymptomatic healthy group
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Grip Strength | Data collection will continue until September 2019. Data analysis and report preparation will be completed by August 2020.
  Grip strenght was examined using a hand dynamometer (Lafayette Proffessional Hand Held Dynamometer, USA).

SECONDARY OUTCOMES:
Two-Point Pinch Strength | Data collection will continue until September 2019. Data analysis and report preparation will be completed by August 2020.
  It was evaluated by pinchmeter (Lafayette,USA).
Three-Point Pinch Strength | Data collection will continue until September 2019. Data analysis and report preparation will be completed by August 2020.
  It was evaluated by pinchmeter (Lafayette,USA).
Lateral Pinch Strength | Data collection will continue until September 2019. Data analysis and report preparation will be completed by August 2020.
  It was evaluated by pinchmeter (Lafayette,USA).
DASH score | Data collection will continue until September 2019. Data analysis and report preparation will be completed by August 2020.
  The DASH score provides information about the general functionality of the upper extremity and especially activities of hand.
Wrist Joint Position Sense | Data collection will continue until September 2019. Data analysis and report preparation will be completed by August 2020.
  Wrist joint position sense was evaluated by goniometric re-position error test ( in 30◦ wrist extansion, 3 repeat ).

CONTACTS AND LOCATIONS:
Overall Officials: İlknur NAZ GÜRŞAN, PhD, Principal Investigator — İzmir Katip Celebi University, Faculty of Health Sciences
Locations (1):
- Izmir Katip Celebi University Ataturk Research and Training Hospital, Izmir, Izmir/ Cigli, Turkey (Türkiye)

REFERENCES:
- [Background] INNES, E. V. Handgrip strength testing: a review of the literature. Australian Occupational Therapy Journal, 1999, 46.3: 120-140.
- [Background] Mathiowetz V, Weber K, Volland G, Kashman N. Reliability and validity of grip and pinch strength evaluations. J Hand Surg Am. 1984 Mar;9(2):222-6. doi: 10.1016/s0363-5023(84)80146-x. PMID 6715829
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Navsarikar A, Gladman DD, Husted JA, Cook RJ. Validity assessment of the disabilities of arm, shoulder, and hand questionnaire (DASH) for patients with psoriatic arthritis. J Rheumatol. 1999 Oct;26(10):2191-4. PMID 10529138
- [Background] Feced Olmos CM, Alvarez-Calderon O, Hervas Marin D, Ivorra Cortes J, Pujol Marco C, Roman Ivorra JA. Relationship between structural damage with loss of strength and functional disability in psoriatic arthritis patients. Clin Biomech (Bristol). 2019 Aug;68:169-174. doi: 10.1016/j.clinbiomech.2019.06.009. Epub 2019 Jun 11. PMID 31220740
- Available data/document: Clinical Study Report — http://ard.bmj.com/content/79/Suppl_1/555.2